CLINICAL TRIAL: NCT04408833
Title: Measurement of Dietary Lipid Oxidation in Toddlers - a Method Study
Brief Title: Palmitate Study: A Method Study of Dietary Lipid Oxidation in Toddlers
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 249922
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to measure how toddlers burn fat after drinking milk that has some fat molecules that can be tracked based on how heavy they are.

DETAILED DESCRIPTION:
The purpose of this research is to measure how toddlers burn fat after drinking milk that has some fat molecules that can be tracked based on how heavy they are. These molecules are not dangerous. By collecting several urine samples throughout a 24-hour window (about 7 urine samples or more) after drinking the fat molecules, we will be able to measure how fast your toddler is sending out (excreting) these samples in the urine. This will tell us how fast your toddler is using fat for energy. This will also help determine the best urine collection schedule for studies using this technology.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male or female
* Toilet trained or not

Exclusion Criteria:

* Diagnosed metabolic disease

Ages: 23 Months to 25 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 10 toddlers approximately two years of age from ongoing studies or as a new participant from the community
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
How toddlers burn fat | 24 hours
  collect urine

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, PhD, Principal Investigator — Arkansas Children's Research Institute
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States